CLINICAL TRIAL: NCT01872624
Title: Bone-marrow Derived Mesenchymal Stromal Cells Associated With One-way Endobronchial Valves in Patients With Pulmonary Emphysema: Safety Study
Brief Title: Safety Study of Bone-marrow Derived Mesenchymal Stromal Cells Associated With Endobronchial Valves in Emphysema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Ministry of Health, Brazil (Other Government); National Research Council, Brazil (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government); Universidade Federal do Rio de Janeiro (Other); Pontifícia Universidade Católica do Paraná (Other)
Responsible Party: Principal Investigator, Hugo Goulart de Oliveira, Associate Professor, Hospital de Clinicas de Porto Alegre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-0150
Record Dates: First submitted 2013-06-05; First posted 2013-06-07 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Pulmonary Emphysema
MeSH Terms: conditions — Pulmonary Emphysema | interventions — Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Valves plus cells (Active Comparator): Bronchoscopy Five patients will be selected to receive bone-marrow derived mesenchymal stromal cells delivered bronchoscopically right before insertion of one-way endobronchial valves.
  Interventions: Procedure: Bronchoscopy
- Valves plus saline (Placebo Comparator): Bronchoscopy Five patients will be selected for treatment with one-way endobronchial valves only, with saline injected prior to valve insertion.
  Interventions: Procedure: Bronchoscopy

INTERVENTIONS:
Procedure: Bronchoscopy — Bronchoscopic delivery of one-way valves and bone-marrow derived mesenchymal stromal cells.

SUMMARY:
The combined use of one-way endobronchial valves and bone-marrow derived mesenchymal stromal cells in patients with severe pulmonary emphysema is safe and will contribute to increase quality of life.

DETAILED DESCRIPTION:
In addition to testing the safety of one-way endobronchial valves combined with bone-marrow derived mesenchymal stromal cells, the study will determine the systemic inflammatory potential of cell therapy measured by C-reactive protein levels (CRP), erythrocyte sedimentation rate (ESR) and complete blood count in peripheral blood. Finally, the study will aim at determining if other markers of inflammatory response and remodeling are modulated by this therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe heterogeneous emphysema (heterogeneity > 15%), with heterogeneity defined as the difference between lobes in the percent area covered by parenchymal density greater than -950 Hounsfield Units.
* Estimation of collateral ventilation based on fissure with integrity ≥ 75%.
* Total lung capacity> 100% predicted.
* Residual volume> 150% predicted.
* Forced expiratory volume at the first minute <45% predicted.
* Diffusing capacity of the lungs for carbon monoxide <45% predicted.
* Optimal medical treatment.
* Limitations in daily physical activities.
* Minimum of 4 months without smoking
* Having family support.
* Stage ≥ 2 in modified Medical Research Council Dyspnea Scale (MMRC).

Exclusion Criteria:

* Homogenous emphysema.
* Presence of collateral ventilation.
* Use of systemic corticosteroids (prednisone> 20mg/day or equivalent).
* Pulmonary or extrapulmonary infection.
* Coronary heart disease and/or severe ventricular dysfunction.
* Significant renal or liver disease.
* Immunosuppressive disease.
* Active smoking.
* Cancer prognosis with survival <2 years.
* Psychosocial problems.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-05; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Absence of lung deficits during the procedure and/or in the 4 months follow-up | 4 months

SECONDARY OUTCOMES:
Quality of Life | 120 days
  St. George Respiratory Questionnaire
Pulmonary function | 120 days
  Spirometry, flow-volume curve, post-bronchodilator test, determination of residual volume, airway resistance by plethysmography, diffusing capacity of the lung for carbon monoxide, and six-minute walk test
Inflammation | 120 days
  Collection of blood samples for determination of C-reactive protein (CRP), erythrocyte

CONTACTS AND LOCATIONS:
Overall Officials: Hugo G Oliveira, MD, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre; Patricia RM Rocco, MD, PhD, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (3):
- Brazil (3):
  - Pontificia Universidade Catolica do Parana, Curitiba, Paraná
  - Universidade Federal do Rio de Janeiro, Rio de Janeiro, Rio de Janeiro
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul

REFERENCES:
- [Background] Abreu SC, Antunes MA, Pelosi P, Morales MM, Rocco PR. Mechanisms of cellular therapy in respiratory diseases. Intensive Care Med. 2011 Sep;37(9):1421-31. doi: 10.1007/s00134-011-2268-3. Epub 2011 Jun 9. PMID 21656291
- [Background] de Oliveira HG, Macedo-Neto AV, John AB, Jungblut S, Prolla JC, Menna-Barreto SS, Fortis EA. Transbronchoscopic pulmonary emphysema treatment: 1-month to 24-month endoscopic follow-up. Chest. 2006 Jul;130(1):190-9. doi: 10.1378/chest.130.1.190. PMID 16840401